CLINICAL TRIAL: NCT02971670
Title: Amendment of Phase 1 Clinical Trial of the BioMed rTSST-1 Variant Vaccine in Healthy Adults
Brief Title: Amendment of rTSST-1 Variant Vaccine Phase 1 Clinical Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biomedizinische Forschungs gmbH (Industry)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BioMed0713 B
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Results first posted 2017-05-08 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Toxic-Shock Syndrome; Sepsis
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Group 1 (Experimental): Treatment: rTSST-1 Variant Candidate Vaccine 3 µg
  Interventions: Biological: rTSST-1 Variant Candidate Vaccine
- Dose Group 2 (Experimental): Treatment: rTSST-1 Variant Candidate Vaccine 10 µg
  Interventions: Biological: rTSST-1 Variant Candidate Vaccine
- Dose Group 3 (Experimental): Treatment: rTSST-1 Variant Candidate Vaccine 30 µg
  Interventions: Biological: rTSST-1 Variant Candidate Vaccine
- Dose Group 0 (Placebo Comparator): Control: Al(OH)3 Adjuvant
  Interventions: Biological: rTSST-1 Variant Candidate Vaccine

INTERVENTIONS:
Biological: rTSST-1 Variant Candidate Vaccine — Immunization either according to their former allocated dose (group 4: 3 µg of candidate vaccine or placebo, group 5: 10 µg of candidate vaccine or placebo, group 6: 30 µg of candidate vaccine or placebo) or 3 µg of candidate vaccine or placebo (groups 1 - 3) from Phase I.

SUMMARY:
Toxic Shock Syndrome (TSS) a severe condition with high morbidity and mortality results from the hosts overwhelming inflammatory response and cytokine storm. Staphylococcal superantigen toxins are the main causative agents. Toxic shock syndrome toxin (TSST-1) being responsible for almost all of menstruation associated and more than 50% of all other cases. There is no specific therapy. The Phase I study BioMed0713 demonstrated the safety and tolerability of the BioMed recombinant toxic shock syndrome toxin (rTSST-1) Variant Vaccine in healthy adults.

The aim of this amendment is to demonstrate prolonged safety of the BioMed rTSST-1 Variant Vaccine and to assess persistence of antibodies generated in participants. The second aim of the study is to assess boosterability of the BioMed rTSST-1 Variant Vaccine.

DETAILED DESCRIPTION:
The BioMed rTSST-1 Variant Vaccine has been developed by Biomedizinische ForschungsgmbH as one component of a polyvalent staphylococcal vaccine for the prevention of toxic shock and hyperimmunization of donors for the production of TSST-1 immunoglobulin.

This is a prospective, single-blinded follow-up study of the safety and immunogenicity of the BioMed rTSST1 Variant Vaccine compared to adjuvant in healthy adults.

All subjects who received 2 doses of 100 ng or more of the rTSST-1 Variant Candidate Vaccine or placebo (Groups 1 - 6) will be followed up in a single-blinded manner for long-term immunogenicity 6 - 15 months after their last (= second) immunization to gain more data about persistence of TSST-1 Ab titer. As this part of the study occurs after unblinding of the study subjects, it is termed Part B (for better discrimination from double-blinded Part A).

All participants will be invited for a blood withdrawal to determine TSST-1 antibodies. Independent of the TSST-1 Ab titer level, subjects will receive one booster immunization either according to their former allocated dose (group 4: 3µg or placebo, group 5: 10 µg or placebo, group 6: 30 µg or placebo) or 3µg or placebo (groups 1 - 3) in the same visit.

Placebo will be administered according to the former allocated dose.

The treated subjects will stay two hours after immunization at the department and will be followed up for 6 months.

Rationale for reduced monitoring after immunization and follow up:

The BioMed rTSST-1 Variant Vaccine demonstrated excellent local and systemic tolerability and safety and an absence of adverse events classified as clinically relevant during the conduct of the study. Therefore no abnormal findings are expected and the monitoring of the vaccinated subjects after immunization is reduced to two hours, there are three follow up visits planned, 24h (+-2 h), 28 days (+-7 days) and 6 months (+-28 days) after booster vaccination.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* 18 - 64 years
* written informed consent
* physical exam: no abnormal findings unless considered irrelevant by the investigator
* uneventful medical history
* females: adequate contraception

Exclusion Criteria:

* pregnancy
* positive virology markers at first screening
* signs and symptoms of relevant autoimmunity

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha M Eibl, MD, Study Director — Biomedizinische ForschungsgmbH

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 0
Started | 13 | 2 | 5 | 3
Completed | 9 | 1 | 4 | 1
Not Completed | 4 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 4 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 0 | Total
Number analyzed (Participants) | 13 | 2 | 5 | 3 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 2 | 5 | 3 | 23
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (10.1) | 45 (18.4) | 28.6 (7.9) | 31.3 (10.7) | 35.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 4 | 3 | 14
  Male | 7 | 1 | 1 | 0 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 13 | 2 | 5 | 3 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety
Description: Clinical observation and clinical laboratory values
Time Frame: through 6 months
Population: Out of 23 Subjects responding, 8 subjects were not interested to continue; 15 subjects were included as PP population.
Measure: Number; unit: participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 0
Number analyzed (Participants) | 9 | 1 | 4 | 1
participants | 7 | 1 | 1 | 0

2. Primary Outcome: Persistence of TSST-1 Antibodies
Description: ELISA IgG against rTSST-1. Persistence of antibody was defined as a >/= 4-fold increase in TSST-1 Ab titer as compared to pre-vaccination values.
Time Frame: 6-15 months after last immunization of Phase I
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 0
Number analyzed (Participants) | 13 | 2 | 5 | 3
Participants | 9 | 2 | 3 | 0

3. Secondary Outcome: Boosterability of BioMed rTSST-1 Variant Vaccine
Description: ELISA IgG against rTSST-1. Boosterability was defined as an increase in TSST-1 Ab titer as compared to antibody titers after second vaccination.
Time Frame: through 6 months after third immunization
Population: Out of 23 Subjects responding, 8 subjects were not interested to continue; 15 subjects were included as PP population.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 0
Number analyzed (Participants) | 9 | 1 | 4 | 1
Participants | 8 | 1 | 4 | 0

ADVERSE EVENTS:
Arm/Group | Dose Group 1 | Dose Group 2 | Dose Group 3 | Dose Group 0
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/1 | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 7/9 | 1/1 | 1/4 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Group 1 (N=9) | Dose Group 2 (N=1) | Dose Group 3 (N=4) | Dose Group 0 (N=1)
Non-drug-related Hospitalization (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hospitalization became necessary subsequently to a radius fracture to surgically remove osteosynthesis material from the left arm.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Group 1 (N=9) | Dose Group 2 (N=1) | Dose Group 3 (N=4) | Dose Group 0 (N=1)
Mild to moderate reactions (General disorders) | 7 | 1 | 1 | 0 — All other adverse events were mild to moderate, with symptoms as in Phase I (NCT02340338), and all were classified as not clinically relevant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No